CLINICAL TRIAL: NCT07232004
Title: A First-in-Human, Phase 1a/b, Single-Dose Study of ABBV-547 to Evaluate the Pharmacokinetics, Immunogenicity, Safety, and Tolerability in Adult Participants and Efficacy in Adult Participants
Brief Title: A Study to Evaluate How the Study Drug Moves Through the Body, Adverse Events, and How the Body Tolerates ABBV-547 Injections
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: M26-058
Record Dates: First submitted 2025-11-14; First posted 2025-11-17 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Healthy Volunteer
Keywords: Healthy Volunteer; ABBV-547

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Group 1: ABBV-547 & Placebo (Experimental): Participants will receive either ABBV-547 or placebo.
  Interventions: Drug: ABBV-547; Drug: ABBV-547 Placebo
- Group 2: ABBV-547 & Placebo (Experimental): Participants will receive either ABBV-547 or placebo.
  Interventions: Drug: ABBV-547; Drug: ABBV-547 Placebo
- Group 3: ABBV-547 & Placebo (Experimental): Participants will receive either ABBV-547 or placebo.
  Interventions: Drug: ABBV-547; Drug: ABBV-547 Placebo
- Group 4: ABBV-547 & Placebo (Experimental): Participants will receive either ABBV-547 or placebo.
  Interventions: Drug: ABBV-547; Drug: ABBV-547 Placebo
- Group 5: ABBV-547 & Placebo (Experimental): Participants will receive either ABBV-547 or placebo.
  Interventions: Drug: ABBV-547; Drug: ABBV-547 Placebo
- Group 6: ABBV-547 & Placebo (Experimental): Participants will receive either ABBV-547 or placebo.
  Interventions: Drug: ABBV-547; Drug: ABBV-547 Placebo

INTERVENTIONS:
Drug: ABBV-547 — Injection
Drug: ABBV-547 Placebo — Injection

SUMMARY:
The purpose of this study is to assess how safe, effective, and tolerable ABBV-547 is in adult participants in the United States and Japan.

There will be 2 parts to this study. In Part 1, participants are placed in one of 3 groups where they will receive ABBV-547 at different doses or placebo. There is a 1 in 4 chance participants will receive placebo. In Part 2, participants are placed in one of 3 groups where they will receive ABBV-547 at different doses or placebo. There is a 1 in 7 chance participants will receive placebo. Approximately 87 adult participants will be enrolled at approximately 21 sites in the United States and Japan.

Participants will be administered one dose of ABBV-547 or placebo.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* A condition of general good health, based upon the results of a medical history, physical examination, vital signs, laboratory profile and a 12-lead electrocardiogram (ECG).
* Part 1: BMI is >= 18.0 to <= 29.9 kg/m^2 after rounding to the tenths decimal at Screening. BMI is calculated as weight in kg divided by the square of height measured in meters.
* Part 2: must have discontinued use of phototherapy (e.g., UVA or UVB) at least 2 weeks prior to the baseline visit (Day 1) and PUVA phototherapy at least 4 weeks prior to the baseline visit (Day 1).

Exclusion Criteria:

* History of any clinically significant sensitivity or allergy to any medication or food.
* Part 2: uses any herbal supplements within the 2-week period prior to study treatment administration.
* Part 2: received any biologics including investigational agents within 2.5 half-lives prior to Baseline.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 87 (Estimated)
Dates: Start 2025-11-24 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) | Up to Approximately Day 365
  An AE is defined as any untoward medical occurrence in a patient or clinical investigation in which a participant is administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (2):
- United States (2):
  - CenExel ACT- Anaheim Clinical Trials /ID# 279612, Anaheim, California
  - Acpru /Id# 278638, Grayslake, Illinois

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M26-058